CLINICAL TRIAL: NCT06722599
Title: Four Cycles Taxane With Trastuzumab and Pertuzumab Neoadjuvant Therapy Among T1c HER2 Positive Patients
Brief Title: Four Cycles Taxane With Trastuzumab and Pertuzumab Neoadjuvant Therapy Among Low Risk HER2 Positive Patients
Acronym: LRNacHER2
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z162
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: HER2-positive Breast Cancer
Keywords: neoadjuvant chemotherapy; De-escalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- four cycles of Taxanes combined with target therapy: Four cycle neoadjuvant therapy with taxanes combined with trastuzumab and pertuzumab

SUMMARY:
Neoadjuvant therapy in the treatment of breast cancer is not only a means of breast conserving surgery, but also a sensitive scheme for patients, in order to reduce the treatment grade, low toxicity and high efficiency. Chemotherapy combined with trastuzumab and pertuzumab is the standard neoadjuvant therapy for HER2 positive breast cancer patients. Paclitaxel plus carboplatin (TCb) is the first choice of chemotherapy recommended by major guidelines; As an alternative, single drug Taxus (T) is also listed as class I recommendation in the latest CSCO guidelines, but the level of evidence is slightly insufficient. In the HER2 positive neoadjuvant therapy population, relatively early and low-risk patients may obtain good curative effect in the treatment of single drug taxane chemotherapy combined with double target therapy.

The project plans to adopt an ambispective cohort study, based on the large sample breast disease cohort database established by the breast center of Peking University People's Hospital, and retrospectively include the HER2 positive breast cancer patients with clinical stage T1c, lymph node negative and receiving Taxanes combined with double target neoadjuvant therapy admitted to the center from January 1, 2019 to December 31, 2024. Patients of the same type were prospectively included from January 1, 2025 to December 31, 2028. Objective to evaluate the efficacy and safety of Taxanes combined with double target neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HER2 positive breast cancer were diagnosed by biopsy in Peking University People's hospital;
2. The clinical stages were T1c, N0, M0;
3. Received treatment in our hospital and had hospitalization records;
4. Has signed and agreed to participate in the PKUPH breast disease cohort study;
5. It is up to the clinician to decide whether to add anthracycline chemotherapy in the adjuvant treatment stage.

Exclusion Criteria:

1. Lack of clinical and pathological data (such as imaging data and pathological data);
2. Patients with metastatic breast cancer or bilateral breast cancer;
3. At the same time, they received anti-tumor therapy in other clinical trials, including endocrine therapy and targeted therapy;
4. Receiving other regimens besides the established neoadjuvant regimens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: T1cN0M0 HER2 positive breast cancer patients who received neoadjuvant chemotherapy based on taxanes combined with target therapy
Sampling Method: Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pathology complete response | 4 months
  Postoperative pathology confirmed that the primary breast lesions and axillary lymph nodes had no residual invasive tumor cells (ypT0/is and ypN0)

SECONDARY OUTCOMES:
Invasive disease free survival | 5 years
  the time from study enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.
Disease free survival | 5 years
  the time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.
Breast cancer specific survival | 5 years
  time from study enrollment to death due to breast cancer.
Overall survival | 5 years
  the time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China